CLINICAL TRIAL: NCT05105386
Title: The Impact of Synergies of Indoor Air Pollutants on Childhood Health and Wellbeing
Acronym: SynAir-Child
Status: Not yet recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, NIKOLAOS G. PAPADOPOULOS, PROFESSOR, National and Kapodistrian University of Athens
Other Study IDs: SEP-210769726
Record Dates: First submitted 2021-09-13; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Pollution; Exposure; Environmental Exposure; Childhood Asthma; Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood samples (optional)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SynAir-Child — Monitor the indoor pollutants and their effect on children well being

SUMMARY:
To quantify health effects of synergizing chemical and biological pollutants in a targeted population setting, i.e., school-aged children. Indoor air pollutants will be monitored within the classrooms with high end sensors. Exposure data from additional sources (outdoor, home, transports) will be obtained. Health outcomes will be assessed prospectively using validated medical procedures and real-time tracking with mobile health (mHealth) equipment and a gamified computer app.

DETAILED DESCRIPTION:
Communication with individual schools and families representing diverse cultural and socioeconomic backgrounds, will be conducted and formal participation consents obtained. The target population will include healthy children and be enriched for children with respiratory allergies and asthma. Provision of instructions, training for participation and baseline assessments of respiratory, immune, and mental health using questionnaires and relevant physiological measurements (e.g spirometry, FeNO), will be performed. Sensors will be positioned and cross-checked for functionality.Health data from the cohort will be monitored by a specifically designed gamified application, as well as by state-of-the-art wearable tracking technology. The app will capture input from the participants at large, while the trackers will accurately, continuously, and remotely, identify personalized patterns of all day activity status, heart rate, oxygen saturation, temperature, blood pressure, sleep, respiratory rate, and mechano-acoustic breathing sounds signatures. Sentinel data will be processed in Work Package 6 and integrated in the SynAir-G autonomous sensing platform.

Children will be prospectively followed-up for a school year. Investigators will regularly visit schools to keep sensors running and collect materials. Real-time tracking will be coupled with regular communication and face-to-face visits for health outcome assessments. Devices will be positioned in selected locations. The cohort will also provide the setting for establishing indoor and outdoor interactions, dose-responses in real life, and health outcome data for integration and synergy analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Students of primary schools aged 8-9 years.
2. The subject and/or legal custodian have the verbal, writing and mental ability to understand the intent and character of the study.
3. Written informed consent from the child's parents/guardian's

Exclusion Criteria:

Unwilling to use the application and follow the procedures of the protocol

Ages: 8 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: Children at this age have the ability to understand the character of the study, to handle the app and the wearables, to successfully perform lung function and airway inflammation measurements (as it has been ascertained in the previous FP7_PreDicta and Horizon_CURE projects), to cooperate with blood sampling, while not being yet subjective to hormonal changes of puberty. Moreover, students at this age mainly attend lessons in the same class, thus exposures in the school environment are considered stable,
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory, mental health | One year
  Questionnaires
Immune health | One year
  RNA Sequency/CRP
Oxidative stress | One year
  DNA damage levels in blood cells
Lung function and | One year
  Spirometry
Airway inflammation | One year
  Exhaled nitric oxide
Exhaled volatile compounds | One year
  Breath biopsy
Cardiovascular metrics | One year
  Wearables
Height and weight | One year
  Height in cm and weight in kg will be combined to report BMI (kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: NIKOLAOS G PAPADOPOULOS, Professor, Study Chair — National and Kapodistrian Univeristy of Athens

IPD SHARING:
Plan to Share IPD: Undecided